CLINICAL TRIAL: NCT04972617
Title: Characterization of the Efficacy of Furosemide Depending on Albumin Function - a Prospective Monocentric Observational Study
Brief Title: Characterization of the Efficacy of Furosemide Depending on Albumin Function
Status: Completed | Type: Observational
Sponsor: University of Rostock (Other)
Responsible Party: Principal Investigator, Gerd Klinkmann, Principal Investigator, University of Rostock
Other Study IDs: Albumin - Furosemid
Record Dates: First submitted 2021-07-01; First posted 2021-07-22 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Acute Renal Failure; Critical Illness
Keywords: furosemide; albumin function; albumin
MeSH Terms: conditions — Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- observational group: In patients with intravenous furosemide administration, an additional 15 ml of blood is taken for the analysis of specific parameters as part of the blood sampling necessary for the treatment of the patient.
  The effect of furosemide is assessed on the basis of the patient's urine excretion. For this purpose, fluid intake and excretion are balanced over 6 hours. The blood sample is taken at the beginning of the balancing period.
  In addition, the albumin concentration, ABiC, as well as the total and free concentration of furosemide in the collected urine are determined.
  Interventions: Diagnostic Test: albumin function analysis (ABIC)

INTERVENTIONS:
Diagnostic Test: albumin function analysis (ABIC) — After centrifugation (10 minutes at 4000 rpm), the plasma is aliquoted and stored at minus 80° C until further analysis. The free as well as the total furosemide concentration is determined by HPLC. In addition to the characterisation of the albumin function by means of the ABiC, these samples can also be used for the determination of the albumin concentration (prerequisite for the determination of the ABiC) and free furosemide concentration as well as for the determination of further parameters relevant for the albumin function.
  Other Names: analysis of total furosemide concentration

SUMMARY:
During this prospective, uncontrolled and non-interventional observational study, the influence of albumin function on the efficacy of furosemide will be investigated. The aim of the study is to provide information on the efficacy of furosemide depending on albumin function.

DETAILED DESCRIPTION:
In patients with intravenous furosemide administration, an additional 15 ml of blood is taken for the analysis of specific parameters as part of the blood sampling necessary for the treatment of the patient.

The effect of furosemide is assessed on the basis of the patient's urine excretion. For this purpose, fluid intake and excretion are balanced over 6 hours. The blood sample is taken at the beginning of the balancing period.

In addition, the albumin concentration, ABiC, as well as the total and free concentration of furosemide in the collected urine are determined.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent
* Attending intensive care physician intends to prescribe IV furosemide to increase urine output
* Arterial (central venous if applicable) and urinary catheter in situ

Exclusion Criteria:

* Attending intensive care physician intends to prescribe further doses of diuretic medication (including furosemide infusion) within the 6 hours required for fluid collection
* Patients who received intravenous or oral diuretics (including mannitol) in the 6 hours prior to study enrolment
* Patients who have received other medications (e.g. fludrocortisone) known to affect renal sodium or water excretion in the 24 hours prior to study entry
* Patients with uncontrolled hyperglycaemia (plasma glucose >10mmol/L).
* Patients who were receiving renal replacement therapy prior to the start of the study
* Patients with obstructive uropathy, macroscopic haematuria or intra-abdominal hypertension (>20mmHg)
* Age < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: intensive care patients admitted to University Hospital Rostock
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Change in the ratio of urine output to fluid input after initiation of furosemide therapy in correlation to the ABiC | 6 hours post-dose
  Assessment of the ABiC 5 minutes after furosemid administration as well as urine output and fluid input for 6 hours post-dose for every hour
Change of the levels of the patient-specific unbound furosemide fraction in correlation to the ABiC | 5 minutes post-dose
  Assessment of the patient-specific unbound furosemide fraction 5 minutes after furosemid administration

SECONDARY OUTCOMES:
Influence of disease severity on ABiC | 12 hours
  Correlation of clinical parameters of critical ill patients with the ABiC:
  * Comorbidities of the organ subsystems (cardio-pulmonary, abdominal, nephrological, endocrinological)
  * Drug intake
  * Conditions affecting critically ill patients (haemodynamic status, sepsis, ARDS, nutritional status)
Influence of biochemical parameters on ABiC | 12 hours
  Correlation of biochemical parameters of critical ill patients with the ABiC:
  * Hemogram
  * Acid-base balance
  * Organ-specific parameters (kidney, liver, immune system)
  * Albumin
  * Unbound forusemide fraction
  * Urine analysis

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Mitzner, MD, PhD, Study Director — University Hospital Rostock
Locations (1):
- University Hospital Rostock, Rostock, Mecklenburg-Vorpommern, Germany

IPD SHARING:
Plan to Share IPD: Undecided